CLINICAL TRIAL: NCT07181122
Title: Prospective Observational Evaluation of Quality of Life, Functional Status, and Cognitive Outcomes in Patients With Metastatic Hormone-Sensitive Prostate Cancer Undergoing Androgen Receptor Pathway Inhibitor Therapy
Brief Title: Quality of Life, Functional and Cognitive Outcomes in Patients With Metastatic Hormone-Sensitive Prostate Cancer
Acronym: PRO-MIND
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncology Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-0132; AEŞH-EK-2025-0132 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: Prostate cancer; mHSPC; Androgen receptor pathway inhibitors; Abiraterone; Apalutamide; Enzalutamide; Darolutamide; Quality of life; Cognitive function; Fatigue; Depression; Sleep quality; Patient-reported outcomes
MeSH Terms: conditions — Prostatic Neoplasms; Fatigue; Depression; Sleep Initiation and Maintenance Disorders | interventions — Abiraterone Acetate; apalutamide; enzalutamide; darolutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Androgen Receptor Pathway Inhibitor Cohort: Men with metastatic hormone-sensitive prostate cancer receiving androgen receptor pathway inhibitors (abiraterone acetate, apalutamide, enzalutamide, or darolutamide) in combination with standard androgen deprivation therapy. Participants will be assessed at baseline, 3 months, and 6 months for quality of life, cognitive function, fatigue, depression, sleep quality, clinical parameters, and treatment-related adverse events.
  Interventions: Drug: Androgen Receptor Pathway Inhibitors (ARPIs)

INTERVENTIONS:
Drug: Androgen Receptor Pathway Inhibitors (ARPIs) — Men with metastatic hormone-sensitive prostate cancer will receive androgen receptor pathway inhibitors (abiraterone acetate, apalutamide, enzalutamide, or darolutamide) in addition to standard androgen deprivation therapy. The choice of ARPI will be determined by routine clinical practice. The study does not assign treatments; it observes patient outcomes under real-world conditions.
  Other Names: Abiraterone acetate; Apalutamide; Enzalutamide; Darolutamide

SUMMARY:
This prospective observational study will evaluate quality of life, functional status, and cognitive outcomes in men with metastatic hormone-sensitive prostate cancer (mHSPC) receiving androgen receptor pathway inhibitors (ARPIs) in addition to standard androgen deprivation therapy. ARPIs in this study include abiraterone acetate, apalutamide, enzalutamide, and darolutamide, depending on local availability. A total of 102 patients will be enrolled from two academic oncology centers in Türkiye.

Participants will be assessed at baseline, 3 months, and 6 months using validated Turkish versions of established questionnaires: Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog), Functional Assessment of Cancer Therapy-Fatigue (FACT-F), Patient Health Questionnaire-9 (PHQ-9), and Pittsburgh Sleep Quality Index (PSQI). Clinical parameters, ECOG performance status, routine laboratory results, and treatment-related adverse events will also be recorded.

The primary outcomes are longitudinal changes in FACT-Cog and FACT-F scores. Secondary outcomes include changes in depression, sleep quality, laboratory results, and adverse events. This study will provide real-world evidence on how ARPI therapy affects cognitive health and quality of life in patients with mHSPC.

DETAILED DESCRIPTION:
Metastatic hormone-sensitive prostate cancer (mHSPC) is a disease stage in which systemic treatment strategies significantly affect survival, functional status, and quality of life. The incorporation of androgen receptor pathway inhibitors (ARPIs) into clinical practice has improved oncological outcomes, yet their influence on cognitive function, fatigue, mood, and sleep requires further real-world investigation.

In this study, the term androgen receptor pathway inhibitors (ARPIs) refer to abiraterone acetate, apalutamide, enzalutamide, and darolutamide. While abiraterone, apalutamide, and enzalutamide are widely used in routine practice in Türkiye, darolutamide may also be included when accessible. All patients will receive ARPIs in combination with standard androgen deprivation therapy (ADT).

This prospective, multicenter, observational cohort study will enroll 102 patients with newly diagnosed mHSPC at Ankara Etlik City Hospital and Gazi University. Assessments will take place at baseline, 3 months, and 6 months.

Validated Turkish patient-reported outcome instruments will be applied:

FACT-Cog: score range 0-148; higher scores = better cognitive functioning.

FACT-F: score range 0-52; higher scores = less fatigue.

PHQ-9: score range 0-27; cut-offs: 5 (mild), 10 (moderate), 15 (moderately severe), 20+ (severe depression).

PSQI: score range 0-21; global score >5 indicates poor sleep quality.

Additional measures will include ECOG performance status (0-5; higher = worse functioning), demographic and clinical characteristics, comorbidities, and routine laboratory tests. Treatment-related adverse events will be recorded according to CTCAE criteria.

The primary outcomes are longitudinal changes in FACT-Cog and FACT-F scores between baseline, 3 months, and 6 months. Secondary outcomes include changes in PHQ-9 and PSQI scores, ECOG performance status, and laboratory results, as well as adverse event profiles. Exploratory analyses will assess the relationship between clinical or laboratory variables and patient-reported outcomes.

Statistical analyses will include descriptive statistics, group comparisons, and repeated-measures modeling. Multivariable regression will be applied to identify predictors of impaired cognitive or functional outcomes.

By incorporating validated Turkish instruments and explicitly defining ARPI agents, this study aims to generate robust real-world evidence on the cognitive, functional, and quality-of-life effects of ARPI therapy in mHSPC. The findings are expected to guide supportive care strategies and optimize treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically or cytologically confirmed metastatic hormone-sensitive prostate cancer (mHSPC)
* Planned initiation of androgen deprivation therapy (ADT) plus an androgen receptor pathway inhibitor (abiraterone, apalutamide, or enzalutamide) as part of routine clinical care
* Ability to complete patient-reported outcome questionnaires (FACT-Cog, FACT-F, PHQ-9, PSQI)
* Written informed consent obtained

Exclusion Criteria:

* Prior systemic therapy for metastatic prostate cancer (except ≤3 months of ADT)
* Known history of severe cognitive impairment that precludes completion of questionnaires
* Concurrent active malignancy requiring systemic treatment
* Inability to comply with study procedures or follow-up
* Any condition judged by the investigator to compromise participation or data integrity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically male participants are eligible, as prostate cancer occurs exclusively in males. Self-identified gender does not alter eligibility since inclusion is based on biological sex.
Study Population: Male patients aged 18 years and older with histologically or cytologically confirmed metastatic hormone-sensitive prostate cancer, initiating androgen deprivation therapy plus an androgen receptor pathway inhibitor (abiraterone, apalutamide, or enzalutamide) in oncology clinics. Participants will be consecutively enrolled at Ankara Etlik City Hospital and Gazi University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) Total Score | Baseline, 3 months, and 6 months after treatment initiation
  FACT-Cog total score ranges from 0 to 148, with higher scores indicating better cognitive functioning. Both continuous change (follow-up minus baseline) and categorical decline (≥10-point decrease from baseline, indicating clinically meaningful cognitive deterioration) will be assessed.
Change From Baseline in Functional Assessment of Cancer Therapy - Fatigue (FACT-F) Score | Baseline, 3 months, and 6 months after treatment initiation
  FACT-F total score ranges from 0 to 52, with higher scores indicating less fatigue burden (better status). Both continuous change and categorical threshold (FACT-F ≤34 = clinically significant fatigue) will be evaluated.

SECONDARY OUTCOMES:
Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Depression Score | Baseline, 3 months, and 6 months after treatment initiation
  PHQ-9 total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. Both continuous change and categorical threshold (PHQ-9 ≥10 = moderate-to-severe depression) will be reported.
Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Global Score | Baseline, 3 months, and 6 months after treatment initiation
  PSQI global score ranges from 0 to 21, with higher scores indicating poorer sleep quality. Both continuous change and categorical threshold (PSQI >5 = poor sleep quality) will be assessed.
Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline, 3 months, and 6 months after treatment initiation
  ECOG performance status ranges from 0 (fully active) to 4 (completely disabled), with higher scores indicating worse functional status. Both continuous change and categorical threshold (≥1-point worsening = functional decline) will be evaluated.
Change From Baseline in Liver Function Parameters | Baseline, 3 months, and 6 months after treatment initiation
  Change in serum AST (U/L), ALT (U/L), total bilirubin (mg/dL), and alkaline phosphatase (U/L). Higher levels reflect worsening liver function. Continuous values will be reported.
Change From Baseline in Renal Function Parameters | Baseline, 3 months, and 6 months after treatment initiation
  Change in serum creatinine (mg/dL) and estimated glomerular filtration rate (eGFR, mL/min/1.73 m²). Higher creatinine and lower eGFR reflect worse renal function. Continuous values will be reported.
Change From Baseline in Electrolyte Levels | Baseline, 3 months, and 6 months after treatment initiation
  Change in serum sodium, potassium, calcium, and other routine electrolytes (mmol/L). Both increases and decreases outside the normal reference range will be noted. Continuous values will be reported.
Change From Baseline in Complete Blood Count (CBC) | Baseline, 3 months, and 6 months after treatment initiation
  Change in hemoglobin (g/dL), white blood cell count, neutrophils, lymphocytes, and platelet count (×10⁹/L). Both continuous changes and categorical thresholds (e.g., anemia = hemoglobin <12 g/dL) will be reported.

OTHER OUTCOMES:
Incidence of Treatment-Related Adverse Events (CTCAE v5.0) | Baseline to 6 months after treatment initiation
  Number and type of adverse events attributed to androgen receptor pathway inhibitor therapy, graded according to CTCAE v5.0 (Grade 1 = mild to Grade 5 = death, with higher grades indicating greater severity).
Correlation Between Clinical/Laboratory Parameters and Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) Score | Baseline to 6 months
  Exploratory correlation between clinical/laboratory parameters (e.g., metabolic profile, PSA) and FACT-Cog score change. Both continuous scores (range: 0-148; higher scores = better cognitive function) and categorical decline (≥10-point decrease from baseline = meaningful deterioration) will be analyzed.
Correlation Between Clinical/Laboratory Parameters and Functional Assessment of Cancer Therapy - Fatigue (FACT-F) Score | Baseline to 6 months
  Exploratory correlation between clinical/laboratory parameters and FACT-F score change. Both continuous scores (range: 0-52; higher scores = less fatigue burden) and categorical threshold (FACT-F ≤34 = clinically significant fatigue) will be analyzed.
Correlation Between Clinical/Laboratory Parameters and Patient Health Questionnaire-9 (PHQ-9) Depression Score | Baseline to 6 months
  Exploratory correlation between clinical/laboratory parameters and PHQ-9 score change. Both continuous scores (range: 0-27; higher scores = worse depression) and categorical threshold (PHQ-9 ≥10 = moderate-to-severe depression) will be analyzed.
Correlation Between Clinical/Laboratory Parameters and Pittsburgh Sleep Quality Index (PSQI) Global Score | Baseline to 6 months
  Exploratory correlation between clinical/laboratory parameters and PSQI score change. Both continuous scores (range: 0-21; higher scores = poorer sleep quality) and categorical threshold (PSQI >5 = poor sleep quality) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital Medical Oncology Department, Ankara, Yenimahalle
  - Gazi University Medical Oncology Department, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No